CLINICAL TRIAL: NCT07186777
Title: Comparative Predictive Accuracy of EMTRAS, REMS, and GAP Scores for Mortality, Endotracheal Intubation, and Length of Hospitalization in Trauma Patients: The First Prospective Cohort Study From Iraq
Brief Title: Comparison of EMTRAS, REMS, and GAP Scores in Trauma
Acronym: TRAPS
Status: Not yet recruiting | Type: Observational
Sponsor: Al-Nahrain University (Other)
Responsible Party: Principal Investigator, Abdul-Ilah R. Khamis, Principal Investigator, Al-Nahrain University
Other Study IDs: UNCOMIRB2025934
Record Dates: First submitted 2025-09-16; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Trauma Patients
Keywords: EMTRAS; REMS; GAP; Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this prospective multicenter cohort study is to evaluate and compare the predictive utility of the EMTRAS, REMS, and GAP scores in determining key outcomes among trauma patients admitted to participating hospitals in Iraq. The primary outcomes of interest include mortality, the need for endotracheal intubation, and length of hospitalization.

The main questions it aims to answer are:

How accurately do EMTRAS, REMS, and GAP scores predict mortality in trauma patients?

How effective are these scores in predicting the need for endotracheal intubation?

How well do these scores correlate with hospitalization duration in trauma patients?

Participants will:

Be assessed using EMTRAS, REMS, and GAP scores upon admission to the emergency department.

Have their clinical outcomes, including survival, intubation requirements, and length of hospital stay, monitored throughout their hospitalization.

DETAILED DESCRIPTION:
Trauma continues to pose a major global public health challenge, accounting for millions of deaths and disabilities each year, with low and middle income countries bearing a disproportionately high burden . Studies suggest that injuries will rise further among the leading causes of mortality, with road traffic accidents, falls, and suicide being among the most prevalent contributors. Approximately 90 percent of trauma deaths occur in low and middle income settings, and a significant portion of these fatalities are considered preventable with the appropriate care.

Efficient risk stratification plays an important role in managing trauma patients, particularly in emergency settings where delays in treatment can have fatal outcomes. Early identification of severely injured individuals supports timely referral and initiation of interventions, both of which are consistently associated with reduced morbidity and mortality.

A wide range of trauma scoring systems have been developed to estimate injury severity, guide triage decisions, and predict outcomes. Yet many established scores, such as the Injury Severity Score and the Trauma and Injury Severity Score, depend on detailed anatomical information that is often unavailable during the critical early phase of emergency care. Others, such as the Revised Trauma Score, are based on physiological indicators but are more complex and may not fully incorporate factors like age or specific injury types. Similarly, scoring systems such as the Acute Physiology and Chronic Health Evaluation II rely on laboratory values, making them less suitable for rapid use in emergency departments.

This limitation becomes even more evident in low and middle income countries, where resource constraints, limited access to complete medical records, and varying trauma patterns make it difficult to apply many existing scoring tools. The need for simple, reliable, and rapid assessment tools that can be applied at the point of care in these environments is especially urgent.

This study focuses on three trauma scores that can be applied early in a patient's clinical course and require only minimal resources: the Emergency Trauma Score, the Rapid Emergency Medicine Score, and the Glasgow Coma Scale Age Pressure score.

The Emergency Trauma Score was developed to estimate the risk of mortality in adult trauma patients using four parameters: age, Glasgow Coma Scale, base excess, and prothrombin time. These values are typically available within 30 minutes of arrival in the emergency department, and this score does not depend on anatomical injury data, making it suitable for early prognostic assessment. The Rapid Emergency Medicine Score is a simplified version of the Acute Physiology and Chronic Health Evaluation II and includes the Glasgow Coma Scale, respiratory rate, oxygen saturation, mean arterial pressure, heart rate, and age. Although originally developed for patients with non-traumatic conditions this score has demonstrated promising predictive ability in trauma populations as well. A modified version of this score, known as the modified Rapid Emergency Medicine Score, was later created to optimize performance in trauma patients. This version adjusts the weight given to age and the Glasgow Coma Scale and replaces mean arterial pressure with systolic blood pressure. The Glasgow Coma Scale Age Pressure score is derived from the Mechanism Glasgow Coma Scale Age Pressure score by removing the mechanism of injury component. It focuses exclusively on physiological variables, specifically Glasgow Coma Scale, age, and systolic blood pressure. The score can be calculated quickly based on a patient's initial clinical status and vital signs, making it especially well-suited for use in settings with limited resources. Previous studies have shown that it has strong predictive ability for mortality.

Although these trauma scores have demonstrated potential, most validation studies have been conducted in high income countries or through single-center retrospective designs. To increase generalizability and relevance to diverse healthcare environments, there is a need for prospective multicenter research, particularly in settings with limited resources and infrastructure.

This current study presents a multicenter prospective cohort analysis from Iraq, a country facing a substantial burden of trauma and significant healthcare challenges. This research compares the accuracy of the Emergency Trauma Score, Rapid Emergency Medicine Score, and Glasgow Coma Scale Age Pressure score in predicting in-hospital mortality among adult trauma patients. The findings aim to offer evidence-based insights that could improve trauma triage and clinical decision-making in resource-constrained environments.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the emergency department with trauma.
* Patients or their legal guardians must provide informed consent to participate in the study.
* Admission within 12 hours of injury.

Exclusion Criteria:

* Patients with incomplete clinical data or those discharged before scoring can be performed.
* Pregnant patients (due to specific physiological considerations not accounted for by the scoring system).
* Patients who died before arrival or were declared dead on arrival.
* Patients who refuse participation or for whom informed consent cannot be obtained.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of adult trauma patients (≥16 years) admitted to the emergency departments of participating tertiary hospitals in Iraq. Eligible patients will include those with blunt or penetrating trauma who present within 12 hours of injury. Patients will be assessed using EMTRAS, REMS, and GAP scores at admission, with outcomes monitored until discharge or in-hospital death.
Sampling Method: Non-Probability Sample
Enrollment: 188 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Accuracy Assessment of EMTRAS, REMS, and GAP Scores in Predicting In-Hospital Mortality | From admission to hospital discharge or death, up to 30 days.
  This outcome evaluates the ability of EMTRAS (range 0-12), REMS (range 0-26), and GAP (range 3-24) to predict in-hospital mortality among trauma patients. Higher EMTRAS and REMS scores, and lower GAP scores, are expected to correlate with increased mortality risk.

SECONDARY OUTCOMES:
Accuracy Assessment of EMTRAS, REMS, and GAP Scores in Predicting the Need for Endotracheal Intubation | From emergency department admission to intubation, discharge, or in-hospital death (up to 30 days).
  This outcome evaluates the predictive performance of EMTRAS (range 0-12), REMS (range 0-26), and GAP (range 3-24) in identifying trauma patients requiring endotracheal intubation during hospitalization. Higher EMTRAS and REMS scores, and lower GAP scores, are expected to be associated with an increased likelihood of intubation.
Accuracy Assessment of EMTRAS, REMS, and GAP Scores in Predicting Length of Hospitalization | From hospital admission to discharge, up to 30 days.
  This outcome assesses the ability of EMTRAS (range 0-12), REMS (range 0-26), and GAP (range 3-24) to predict hospitalization duration. Patients with lower severity scores (low EMTRAS/REMS or high GAP) are expected to have shorter hospital stays, while those with higher severity scores are likely to require prolonged hospitalization.
Accuracy Assessment of EMTRAS, REMS, and GAP Scores in Predicting In-Hospital Morbidity | From hospital admission to discharge or death, up to 30 days.
  This outcome evaluates the incidence and types of complications (morbidity) experienced by trauma patients, as predicted by EMTRAS (0-12), REMS (0-26), and GAP (3-24) scores. Higher EMTRAS and REMS values, and lower GAP scores, are expected to correlate with increased morbidity, including respiratory complications, infections, prolonged mechanical ventilation, and other trauma-related adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- College of Medicine - Al-Nahrain University, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rehn M, Perel P, Blackhall K, Lossius HM. Prognostic models for the early care of trauma patients: a systematic review. Scand J Trauma Resusc Emerg Med. 2011 Mar 20;19:17. doi: 10.1186/1757-7241-19-17. PMID 21418599
- [Background] WHO Global Health Estimates. INJURIES VIOLENCE THE FACTS.; 2014.https://iris.who.int/bitstream/handle/10665/149798/9789241508018_eng.pdf?sequence=1
- [Background] Whitaker J, O'Donohoe N, Denning M, Poenaru D, Guadagno E, Leather AJM, Davies JI. Assessing trauma care systems in low-income and middle-income countries: a systematic review and evidence synthesis mapping the Three Delays framework to injury health system assessments. BMJ Glob Health. 2021 May;6(5):e004324. doi: 10.1136/bmjgh-2020-004324. PMID 33975885
- [Result] Granstrom A, Schandl A, Martensson J, Strommer L. Using the GAP score as a complement to the NISS score in identifying severely injured patients- A registry-based cohort study of adult trauma patients in Sweden. Injury. 2024 Sep;55(9):111709. doi: 10.1016/j.injury.2024.111709. Epub 2024 Jun 28. PMID 38969590
- [Result] GJRA - Global Journal for Research Analysis - Diagnostic Accuracy of Rapid Emergency Medicine Score (REMS) as a prognostic marker and its comparison with traditional scoring systems in trauma. (n.d.). https://www.worldwidejournals.com/global-journal-for-research-analysis-GJRA/file.php?val=diagnostic-accuracy-of-rapid-emergency-medicine-score-rems-as-a-prognostic-marker-and-its-comparison-with-traditional-scoring-systems-in-trauma_January_2023_7615446958_8010945.pdf
- [Result] Karakus A, Yilmaz S, Demirci S, et al. An evaluation of trauma scores (RTS, GAP, EMTRAS) on mortality in multiple trauma patients. J Emerg Med. 2023;65(1):1-8. doi:10.1016/j.jemermed.2023.04.012
- [Result] Phunghassaporn N, Sukhvibul P, Techapongsatorn S, Tansawet A. Accuracy and external validation of the modified rapid emergency medicine score in road traffic injuries in a Bangkok level I trauma center. Heliyon. 2022 Dec 10;8(12):e12225. doi: 10.1016/j.heliyon.2022.e12225. eCollection 2022 Dec. PMID 36568674
- [Result] Joosse P, de Jong WJ, Reitsma JB, Wendt KW, Schep NW, Goslings JC. External validation of the Emergency Trauma Score for early prediction of mortality in trauma patients. Crit Care Med. 2014 Jan;42(1):83-9. doi: 10.1097/CCM.0b013e31829e53f5. PMID 23982027
- [Result] Mangini, M., Di Valvasone, S., Greco, C., Ognibene, A., Cappuccini, G., Spina, R., Tartaglia, R., Zagli, G., & Peris, A. (2010). Validation of the new proposed Emergency Trauma Score (EMTRAS). Critical Care, 14(Suppl 1), P252. https://doi.org/10.1186/cc8484
- [Result] Kumar, G., Kaur, R., Yadav, R., & Kachru, N. (2022). Comparison of Emergency Trauma Score (EMTRAS) with Rapid Emergency Medicine Score (REMS) for Prediction of Early Mortality in Adult Trauma Patients. Archives of Anesthesia and Critical Care. https://doi.org/10.18502/aacc.v8i3.9608
- [Result] Park HO, Kim JW, Kim SH, Moon SH, Byun JH, Kim KN, Yang JH, Lee CE, Jang IS, Kang DH, Kim SC, Kang C, Choi JY. Usability verification of the Emergency Trauma Score (EMTRAS) and Rapid Emergency Medicine Score (REMS) in patients with trauma: A retrospective cohort study. Medicine (Baltimore). 2017 Nov;96(44):e8449. doi: 10.1097/MD.0000000000008449. PMID 29095289
- [Result] Imhoff BF, Thompson NJ, Hastings MA, Nazir N, Moncure M, Cannon CM. Rapid Emergency Medicine Score (REMS) in the trauma population: a retrospective study. BMJ Open. 2014 May 2;4(5):e004738. doi: 10.1136/bmjopen-2013-004738. PMID 24793256
- [Result] Miller RT, Nazir N, McDonald T, Cannon CM. The modified rapid emergency medicine score: A novel trauma triage tool to predict in-hospital mortality. Injury. 2017 Sep;48(9):1870-1877. doi: 10.1016/j.injury.2017.04.048. Epub 2017 Apr 25. PMID 28465003
- [Result] Olsson T, Terent A, Lind L. Rapid Emergency Medicine score: a new prognostic tool for in-hospital mortality in nonsurgical emergency department patients. J Intern Med. 2004 May;255(5):579-87. doi: 10.1111/j.1365-2796.2004.01321.x. PMID 15078500
- [Result] Kumar G, Kaur R, Yadav R, Kachru N. Comparison of Emergency Trauma Score (EMTRAS) with Rapid Emergency Medicine Score (REMS) for prediction of early mortality in adult trauma patients. Arch Anesthesiol Crit Care. 2022;8(3):193-200.
- [Result] Ahun E, Koksal O, Sigirli D, Torun G, Donmez SS, Armagan E. Value of the Glasgow coma scale, age, and arterial blood pressure score for predicting the mortality of major trauma patients presenting to the emergency department. Ulus Travma Acil Cerrahi Derg. 2014 Jul;20(4):241-7. doi: 10.5505/tjtes.2014.76399. PMID 25135017
- [Result] Mohammed S, Ali Y, Hasan M, et al. Trauma care in Iraq: challenges and opportunities. BMC Emerg Med. 2022;22:90. doi:10.1186/s12873-022-00653-1